CLINICAL TRIAL: NCT02656459
Title: Longitudinal Gene Expression Profiling in Adults After Traumatic Injury
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-35447
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Sepsis; Trauma; Infection
Keywords: gene expression
MeSH Terms: conditions — Sepsis; Wounds and Injuries; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood RNA specimens will be retained up to 3 years after study end.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 11-gene set — This trial is NOT interventional. The 11-gene set / Sepsis MetaScore will be tested post-hoc.
  Other Names: Sepsis MetaScore

SUMMARY:
The purpose of this study is to examine the immune response to traumatic injury and subsequent infections in critically ill adults. Traumatic injuries lead to severe dysregulation of the immune system, and predispose to severe infections. Diagnosing these infections in a timely manner is paramount in reducing morbidity and mortality, but diagnosis is made difficult by the inflammatory response to trauma. The main purpose of the study is to prospectively test the diagnostic power of the expression of an 11-gene set which the investigators recently published (Sweeney et al., Sci Transl Med, 2015). Since the timing of an acquired infection cannot be determined a priori, this study is designed to be a longitudinal examination of a cohort of traumatically injured adults. The investigators will draw blood at regular intervals, as well as at day of diagnosis of infection for any patient that are diagnosed with an infection. The investigators will then assay the blood for gene expression levels post hoc, and correlate the molecular profiles with clinical information to establish a prospective estimate of diagnostic power.

DETAILED DESCRIPTION:
Consecutive patients who meet criteria (see below) will be enrolled. Whole blood will be drawn and stored in PAXgene tubes. Blood will be drawn within 24 hours of ICU admission (ICU day 1), and then every three days subsequently (ICU days 4, 7, 10, 13) for two weeks. In addition, a tube of blood will be drawn at the time of clinical diagnosis of infection, if an infection is diagnosed (see below). Patients who are discharged from the ICU prior to two weeks will no longer be profiled. The hour and date of admission, and the hour and date of each subsequent blood draw, will be recorded.

Rates of hospital-acquired infection after severe traumatic injury run around 30-50%. The investigators will enroll 50 patients, which should net around 20 patients with infections, and 30 time-matched non-infected controls. In total, an average of 4 samples/patient, or 200 total blood samples, are expected.

Diagnosis of Infection:

The main purpose of the study is to examine gene expression response to infections. As a result, careful attention must be paid to how infections are classified. First, two systemic inflammatory reaction syndrome (SIRS) criteria are NOT necessary to be designated as infected. Second, the time of diagnosis of infection (and the time of extra blood sampling) will be the time of clinical diagnosis, not the later time that cultures turn positive. It will thus be based on clinical judgement. Finally, post-hoc criteria for infections are described elsewhere. Patients need to eventually meet these criteria to be counted as infected; this will be done in the analysis phase, not the clinical phase.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adults (>=18 years old) admitted to the ICU after blunt traumatic injury.

Exclusion Criteria:

* Patients with isolated traumatic head or spinal cord injuries will not be included.
* Furthermore, patients with prior or under continuous antibiotic therapy will be excluded (e.g. in case of intestinal perforation).
* We will not exclude patients who are given <=24 hours of perioperative antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No patients will be enrolled at Stanford. All enrollment will be done at Universitätsmedizin Göttingen. ICU admissions will be reviewed by the local research team; all patients admitted for blunt trauma will then be screened by chart review for matching inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
11-gene set / Sepsis MetaScore | Patients with infections will be compared to time-matched patients without infections (+/- 24 hours).
  Time-matched controls are necessary to prevent bias due to changes over time that occur with recovery from injury.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E Sweeney, MD, PhD, Principal Investigator — Stanford University; Purvesh Khatri, PhD, Principal Investigator — Stanford University
Locations (3):
- Stanford University, Stanford, California, United States
- Germany (2):
  - University Hospital Essen, Essen
  - University of Gottigen, Göttingen

REFERENCES:
- [Background] Sweeney TE, Shidham A, Wong HR, Khatri P. A comprehensive time-course-based multicohort analysis of sepsis and sterile inflammation reveals a robust diagnostic gene set. Sci Transl Med. 2015 May 13;7(287):287ra71. doi: 10.1126/scitranslmed.aaa5993. PMID 25972003
- [Background] Sweeney TE, Khatri P. Comprehensive Validation of the FAIM3:PLAC8 Ratio in Time-matched Public Gene Expression Data. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1260-1. doi: 10.1164/rccm.201507-1321LE. No abstract available. PMID 26568247